CLINICAL TRIAL: NCT01532063
Title: Risk Factors of Difficult Intubation and Related Complications in Adults in Intensive Care Units(ICU)
Brief Title: Risk Factors of Difficult Intubation and Related Complications in Adults in Intensive Care Units: FRIDA-Rea
Acronym: FRIDA-Rea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8819; 2012-A00651-42 (Other: RCB number)
Record Dates: First submitted 2012-02-08; First posted 2012-02-13 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Difficult Intubation
Keywords: Difficult intubation; Intensive care units; Risk factors; Incidence; Complications; Intubation in Intensive Care Unit; More than 2 attempts of intubation; Intubation attempts lasting more than 10 minutes
MeSH Terms: interventions — Intubation; Intensive Care Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INTUBATION (Other): Subjects intubed in Intensive Care Unit
  Interventions: Procedure: INTUBATION IN INTENSIVE CARE UNIT

INTERVENTIONS:
Procedure: INTUBATION IN INTENSIVE CARE UNIT — Standard intubation procedure used in Intensive Care Unit

SUMMARY:
Difficult intubation is challenging in intensive care units. There are limited data regarding risk factors of difficult intubation in ICU. The primary purpose of the investigators study is to assess the risk factors of difficult airway in adults in ICU.

DETAILED DESCRIPTION:
PURPOSE: Intubation in ICU strongly differs from intubation in operative rooms. The results of studies about risk factors of difficult intubation performed in operative rooms cannot therefore be extrapolated directly to ICU.

The primary purpose of this trial (cf Part "Design" of this registration) is "other" and more particularly "Prognosis" because it is is an assessment of risk factors of difficult airway in intensive care units.

DESIGN AND METHODOLOGY: This is an open prospective multicentric study of intubation in ICU in more than 50 centres. Consecutive intubations will be included in each centre, in order to reach the sample size required (at least 1000 procedures intubations). The usual risk factors of difficult intubation in operative rooms, the demographic parameters and the complications of intubation will be assessed, as well as survival status at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* More or equal to 18 years old
* Men and women
* Informed patient
* Affiliated or benefit from an disease insurance
* Available for a 28 days follow-up
* Intubated patients in Intensive Care Unit

Exclusion Criteria:

* Law protected patients
* Opposed to participate to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difficult intubation | until to 10 minutes
  According to ASA criteria, difficult intubation is measured by attempts lasting more than 10 min or more than two attempts

SECONDARY OUTCOMES:
Complications of intubation in ICU | up to one hour after intubation
  * Respiratory (inhalation, oesophageal intubation, SpO2<80%)
  * Hemodynamic(SAP<65 mm Hg, elevated or low cardiac frequency,rythm troubles, heart attack),
  * Neurologic (agitation),
  * Local (dental trauma, laryngal trauma),
  * Death
  * Complications occuring during one hour after intubation: respiratory (major desaturation: SpO2<80%, pneumothorax, persistent hypoxia with SpO2<80%), hemodynamic (persistent hypotension: SAP<90 mm Hg despite of vascular filling, rythm troubles, heart attack, introduction or majoration of amines posology), neurologic(agitation), death
Mortality at 28 days after difficult intubation | up to 28 days after difficult intubation
  Survival status at Day 28 or date of death if patient dead before.
Incidence of difficult intubation in ICU | up to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Samir SJ JABER, MD,PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Saint Eloi, Montpellier, France

REFERENCES:
- [Derived] Perbet S, De Jong A, Delmas J, Futier E, Pereira B, Jaber S, Constantin JM. Incidence of and risk factors for severe cardiovascular collapse after endotracheal intubation in the ICU: a multicenter observational study. Crit Care. 2015 Jun 18;19(1):257. doi: 10.1186/s13054-015-0975-9. PMID 26084896
- [Derived] De Jong A, Molinari N, Pouzeratte Y, Verzilli D, Chanques G, Jung B, Futier E, Perrigault PF, Colson P, Capdevila X, Jaber S. Difficult intubation in obese patients: incidence, risk factors, and complications in the operating theatre and in intensive care units. Br J Anaesth. 2015 Feb;114(2):297-306. doi: 10.1093/bja/aeu373. Epub 2014 Nov 27. PMID 25431308
- [Derived] De Jong A, Molinari N, Terzi N, Mongardon N, Arnal JM, Guitton C, Allaouchiche B, Paugam-Burtz C, Constantin JM, Lefrant JY, Leone M, Papazian L, Asehnoune K, Maziers N, Azoulay E, Pradel G, Jung B, Jaber S; AzuRea Network for the Frida-Rea Study Group. Early identification of patients at risk for difficult intubation in the intensive care unit: development and validation of the MACOCHA score in a multicenter cohort study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):832-9. doi: 10.1164/rccm.201210-1851OC. PMID 23348979